CLINICAL TRIAL: NCT02284542
Title: NAPS (Non-awake Versus Awake Placement of Spinal Cord Stimulators) Study for the Evaluation of Awake and Non-awake Methods of SCS Paddle Lead Placement
Brief Title: NAPS: Non-awake Versus Awake Placement of Spinal Cord Stimulators
Acronym: NAPS
Status: Completed | Type: Observational
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014-81
Record Dates: First submitted 2014-10-27; First posted 2014-11-06 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Chronic Pain; Sciatica; Failed Back Surgery Syndrome
MeSH Terms: conditions — Chronic Pain; Sciatica; Failed Back Surgery Syndrome | interventions — Wake protein, Drosophila

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with successful trial implant: Patients who have had a successful SCS trial and are indicated for permanent implantation will be approached to participate in this study prior to permanent implantation. Patients will be recruited and enrolled by physicians at any one of the involved sites. Each Investigator will only use one method (awake or non-awake) according to his/her typical practice. Patients will receive treatment from their enrolling physician.
  Interventions: Procedure: Awake; Procedure: Non-Awake

INTERVENTIONS:
Procedure: Awake — Upon approximate lead positioning, the patient is brought to a conscious sedated state while maintaining local anesthetic. Stimulation of the spinal cord through the paddle lead is accomplished with an external pulse generator, while communicating with the patient regarding paresthesia coverage of painful regions.
Procedure: Non-Awake — The patient is maintained under general anesthesia for the full duration of the implant. Upon approximate lead positioning, bilateral EMG of myotomes overlapping dermatomal regions of pain are monitored. Stimulation is delivered through the lead by an external pulse generator in order to elicit compound muscle action potentials (CMAPs) in the target regions. Lead placement is targeted to have symmetric CMAPs (i.e. physiologic midline) and adequate coverage of the painful regions as described by Falowski et al.
  (Falowski et al., 2011).

SUMMARY:
The primary objective is to demonstrate the safety and efficacy of a non-awake implantation method (EMG neuromonitoring) of a SCS paddle lead as compared to an awake implantation method (with local anesthesia and patient feedback).This is a post-market, prospective, multicenter, parallel designed, non-randomized, non-blinded, 6-month study. A minimum of 50 patients will be implanted from up to 4 active sites, coordinated by a single lead investigator.

Patients who have had a successful SCS trial and are indicated for permanent implantation will be approached to participate in this study prior to permanent implantation. Patients will be recruited and enrolled by physicians at any one of the involved sites. Each Investigator will only use one method (awake or non-awake) according to his/her typical practice. Patients will receive treatment from their enrolling physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a successful spinal cord stimulation trial and are indicated for permanent implantation at a participating facility.
* Sign informed consent

Exclusion Criteria:

* < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had a successful SCS trial and are indicated for permanent implantation will be approached to participate in this study prior to permanent implantation. Patients will be recruited and enrolled by physicians at any one of the involved sites. Each Investigator will only use one method (awake or non-awake) according to his/her typical practice. Patients will receive treatment from their enrolling physician.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-11-01; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Safety assessed by the number of adverse events | 24 weeks
Efficacy assessed by the procedure time and number of revision differences between the Awake and Non-Awake methods | 24 weeks

SECONDARY OUTCOMES:
Pain Evaluation | 24 weeks
Pain Location | 24 weeks
Paresthesia assessed by patient reports of tingling, tickling, or prickling sensation | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Falowski, MD, Principal Investigator — Principal Investigator
Locations (4):
- United States (4):
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Neurosciences Institute, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
SJM and Dr. Falowski will share results upon study completion.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-09-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT02284542/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT02284542/ICF_001.pdf